CLINICAL TRIAL: NCT05037864
Title: A Comparison of Posture, Balance and Flexibility in Between Adolescent Ballet Dancers and Sedentary Individuals
Status: Completed | Type: Observational
Sponsor: Irem Kurt (Other)
Responsible Party: Sponsor-Investigator, Irem Kurt, Principal Investigator, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Other Study IDs: IUC3
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Healthy
Keywords: Ballet; Adolescent; Posture; Balance; Flexibility; Physical activity; Dance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ballet Dancer Group (Adolescent Ballet Dancers): Adolescent ballet dancer student aged 7-17 years who have been actively attending a ballet dance school for at least 1 year will be form ballet dancer group. The age, body weight (kg) and height (centimeter) of each individual included in the study will record. The assessment form, which includes demographic data such as, ballet duration(min/day), frequency (times/week) and continuity (year) will record by asking the parents. All measurements will be take before lesson and without warm-up. All measurements will be evaluate by an experienced physiotherapist. Postural alignment will assess with New York Posture Rating Scale (NYPR). Static and dynamic balance will determine with Romberg's Test, Flamingo Balance Test (FBT) and Star Excursion Balance Test (SEBT). Participants will be evaluate for flexibility outcomes by applying following test: sit up and reach test, Thomas test and straight leg raise test. Quality of life will be assess with SF36.
- Control Group (Sedentary Adolescents): The control group (Sedentary Adolescent) of the study, are not ballet dance students who aged 7-17 years and have not experience in competitive sport or activity. The age, body weight (kg) and height (centimeter) of each individual included in the study will record. All measurements will be take before lesson and without warm-up. All measurements will be evaluate by an experienced physiotherapist. Postural alignment will assess with New York Posture Rating Scale (NYPR). Static and dynamic balance will determine with Romberg's Test, Flamingo Balance Test (FBT) and Star Excursion Balance Test (SEBT). Participants will be evaluate for flexibility outcomes by applying following test: sit up and reach test, Thomas test and straight leg raise test. Quality of life will be assess with SF36.

SUMMARY:
Ballet dance are typical specific movement which require balance ability and postural control. Ballet dancers use specific balance exercises. It can be expected, that dancers have an advanced sense of awareness for the placement and motion of their bodies. The effect of ballet dancing on adolescents is still unclear. Therefore, the aim of this study is to determine whether ballet dance has an effect on balance, posture and flexibility in adolescents.

DETAILED DESCRIPTION:
Ballet is as a superlative combination of art and sport that requires high demands musculoskeletal conditioning which works on the development of coordination, balance and associated with efficient strength and flexibility. Balance is a key skill for dance performance for dancers especially for ballet. Ballet dancers use specific balance exercises. It can be expected, that dancers have an advanced sense of awareness for the placement and motion of their bodies. The support surfaces are variable in ballet training, this may also be the reason dancers can better use the information from the somatosensory and vestibular systems. It could be assumed that the effect of ballet training will have a positive effect on postural stability in standing. Postural balance is the act of achieving, maintaining or restoring a state of balance during any posture or activity. It is still unclear whether balance, flexibility and posture in adolescent ballet dancers is different than sedentary adolescent. Therefore, the aim of this study was to assess whether there are differences in balance between adolescent ballet dancers and sedentary adolescent and if these differences are associated with the flexibility and posture. To compare the postural balance between both groups the unipedal standing was chosen, which reduces the quantity of useful and accurate somatosensory information available to the postural control system. Posture analysis and flexibility tests were performed in both groups to compare flexibility and posture on balance. We purpose to compare balance parameters, posture and health quality parameters in adolescent ballet dancers and sedentary adolescent groups.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 7-17 years
* Volunteer
* Does not have any cognitive, mental and psychological problems,
* Does not have any systemic diseases such as rheumatoid arthritis,
* Does not have any neurological problems,
* Additionally, the criteria for the ballet dancers included more than 1 years of ballet experience, and for sedentary they included no experience in competitive sport or activity.

Exclusion Criteria:

* Having severe neurological, visual and auditory problems that may prevent the application of assessment parameters
* Children and their families who cannot obtain written consent from their families.
* Having communication problems

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy adolescent ballet dancers and sedentary individuals
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-10-02 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-07-02 (Actual)

PRIMARY OUTCOMES:
New York Posture Rating Scale (NYPR) | Baseline
  The NYPR applies a quantitative approach to assess proper and improper alignment of various body segments for an individual in the anatomical position. The NYPR published in 1958 includes a set of three figure drawings for each of 13 body alignment segments contributing to overall postural alignment. The 13 body alignment segments include posterior views of the head, shoulders, spine, hip, feet, and arches, and lateral (left side) views of the neck, chest, shoulders, upper back, trunk, abdomen, and lower back. Short verbal descriptions are provided to indicate the visual cues to use as criteria in deciding the score. In this original version, each body segment was scored 5 (correct posture), 3 (slight deviation), or 1 (pronounced deviation). The standard evaluation criteria developed for this test were determined as "very good" if the total score was ≥45, "good" if 40-44, "moderate" if 30-39, "poor" if 20-29 and "bad" if ≤19.
Single leg stance test (SLS) | Baseline
  SLS test is used to assess static balance control. Participants will be asked to stand on a hard floor, on one leg without using any assistive devices, and without support from any surface. SLS times of the participants will be recorded in seconds with the stopwatch and the test will be repeated for both feet.
Flamingo Balance Test (FBT) | Baseline
  The FBT indicates static balance that is simplicity, low cost and it is capable for mass investigations. In this test the participant is standing on his preferred foot, bends his free leg backwards and grips the back of the foot with hand on the same side, standing like a flamingo. The measurement time was kept for one minute. The electronic chronometer was stopped as soon as the participant lost balance or touched the ground. The balance was restored and the electronic chronometer was continued until one minute has passed. Score: Attempts to keep balance within one minute were recorded.
Modified Star Excursion Balance Test (Y-Balance Test) (MSEBT) | Baseline
  The MSEBT is a screening tool commonly used to evaluate lower extremity dynamic stability, neuromuscular control, and injury risk in athletes. It is also used to monitor rehabilitation progress after injury. The SEBT is performed by having the participant stand on one leg and extend the other leg away from their body in eight different directions.
The Short Form health survey with 36 questions (SF-36) | Baseline
  SF-36 is a well-documented scoring system that has been widely used and validated as a quality of life assessment tool for the general population. Multi-item scales have been developed to represent aspects of the following eight physical and mental health domains: Physical Functioning (PF), Role Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role Emotional (RE), and Mental Health (MH). Its most obvious superiority is measuring physical function and related abilities. Subscales evaluate health between 0 and 100, and 0 indicates "bad health", 100 indicates "good health"[9].
Thomas Test | Baseline
  The Thomas Test (also known as Iliacus Test or Iliopsoas Test) is used to measure the flexibility of the hip flexors, which includes the iliopsoas muscle group, the rectus femoris, pectineus, gracillis as well as the tensor fascia latae and the sartorius.The patient should be supine on the examination table, maximally flex both knees, using both arms to ensure that the lumbar spine is flexed and flat on the table and avoids an anterior tilt of the pelvis.The patient then lowers the tested limb toward the table, whilst the contralateral hip and knee is still held in maximal flexion to stabilize the pelvis and flatten out the lumbar lordosis. The length of the iliopsoas is measured by the angle of the hip flexion.
Sit and Reach Test | Baseline
  The Sit and reach test is one of the linear flexibility tests which helps to measure the extensibility of the hamstrings and lower back. Clients/Patients should perform a short warm-up prior to this test with some gentle stretches. The participant's shoes should be removed. A yardstick is placed on the floor and tape is placed across it at a right angle to the 15 inches mark. The client/patient sits with the yardstick between the legs, with the legs extended at right angles to the taped line on the floor. Heels of the feet should touch the edge of the taped line and be about 10 to 12 inches apart.The client/patient should slowly reach forward with extended arms, placing one hand on top of the other facing palms down, as far as possible, holding this position for approximately 2 seconds. The score is the most distant point (cm or in) reached with the fingertips. The best of three trials should be recorded.
Active Straight Leg Raise Test (SLR) | Baseline
  The Straight Leg Raise (SLR) is the most commonly used test, which can be carried out either passively or actively. During the passive SLR (PSLR), the athlete lays supine while one tester moves the lower limb to be tested in hip flexion with the knee fully extended and the ankle relaxed. A second tester measures hamstring flexibility with either a goniometer or an inclinometer, and a third tester might be needed to stabilize the pelvis and the non-tested limb. This test is reliable in assessing hamstring flexibility.

CONTACTS AND LOCATIONS:
Locations (1):
- İrem Kurt, Istanbul, Turkey (Türkiye)